CLINICAL TRIAL: NCT02527148
Title: A Prospective, Randomized, Controlled Trial of Mechanical Axis vs Kinematic Alignment in TKR - With a Follow-up, Longitudinal Study of the Clinical and Radiographic Outcomes
Brief Title: A Trial of Mechanical Axis vs Kinematic Alignment in Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker South Pacific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShapeNZRCT-10
Record Dates: First submitted 2015-08-03; First posted 2015-08-18 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Arthroplasties; Knee Replacement
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OtisMed® ShapeMatch® with Triathlon (Active Comparator): Participants randomised to the Intervention Group will undergo Total Knee Replacement (TKR) with the Stryker Triathlon® Total Knee System and OtisMed® ShapeMatch® Technology with the goal of kinematic alignment (re-aligning the limb to its pre-disease kinematic alignment).
  Interventions: Device: OtisMed® ShapeMatch® Technology; Procedure: Total Knee Replacement; Device: Stryker Triathlon® Total Knee System
- Stryker Precision Knee Navigation (Active Comparator): Participants randomised to the Control Group will undergo Total Knee Replacement (TKR) with the Stryker Triathlon® Total Knee System guided by Stryker Precision Knee Navigation with the goal of neutral alignment to the mechanical axis. This is the standard method for TKR with Triathlon® Knee System and this group will serve as a control reference for the intervention group.
  Interventions: Device: Stryker Precision Knee Navigation; Procedure: Total Knee Replacement; Device: Stryker Triathlon® Total Knee System

INTERVENTIONS:
Device: OtisMed® ShapeMatch® Technology — The appropriate Stryker ShapeMatch® Cutting Guides will be used to guide the surgeons bone resections. The surgeon will implant the knee prostheses following the surgical protocol for Triathlon® Knee System with OtisMed® ShapeMatch® Technology
  Arms: OtisMed® ShapeMatch® with Triathlon
Device: Stryker Precision Knee Navigation — Stryker PrecisioN Knee (4.0) Navigation System, comprising of computer hardware and software and associated instrumentation, will be used for intra-operative alignment and orientation of implant. Navigation trackers will be secured to the femur and tibia and registration of the limb will be undertaken according to the PrecisioN Knee System surgical technique.Femoral and tibial resections, followed by device implantation, will be performed according to the Triathlon Knee System Surgical Protocol.
  Arms: Stryker Precision Knee Navigation
Procedure: Total Knee Replacement
Device: Stryker Triathlon® Total Knee System — Prosthetic components to be implanted including
  * Triathlon® Cruciate Retaining (CR) Total Knee System (cemented), including Femoral Component and Primary Tibial Baseplate;
  * Triathlon® Cruciate Substituting (CS) X3® polyethylene insert;
  * Triathlon® X3 Patella (asymmetric) - treated selectively by surgeon.

SUMMARY:
This is a prospective, randomized, longitudinal study of the clinical outcomes of osteoarthritis patients treated by two different alignment philosophies for total knee replacement. In this study ShapeMatch® cutting guides will be compared to the conventional approach.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or non-pregnant female between the ages of 40-80 years.
* The patient requires a primary total knee replacement and is indicated for computer-assisted surgery.
* Patient is deemed appropriate for a cruciate retaining knee replacement.
* The patient has a primary diagnosis of osteoarthritis (OA).
* The patient has intact collateral ligaments.
* The patient is able to undergo MRI scanning of the affected limb.
* The patient has signed the study specific, ethics-approved, Informed Consent document.
* The patient is willing and able to comply with the specified pre-operative and post-operative clinical and radiographic evaluations.

Exclusion Criteria:

* The patient has a history of total, unicompartmental reconstruction or fusion of the affected joint.
* Patient has had a previous osteotomy around the knee.
* The patient is morbidly obese (BMI ≥ 40).
* The patient has a deformity which will require the use of stems, wedges or augments in conjunction with the Triathlon Total Knee System.
* The patient has a varus/valgus malalignment ≥ 15° (relative to mechanical axis).
* The patient has a fixed flexion deformity ≥ 15°.
* The patient has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* The patient has a systemic or metabolic disorder leading to progressive bone deterioration.
* The patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements.
* Patient has a cognitive impairment, an intellectual disability or a mental illness.
* The patient is pregnant.
* The patient has metal hardware present in the region of the hip, knee or ankle (as this is known to create geometrical distortion in the region of the implant).
* The patient has any known contraindications for undergoing assessment by MRI (e.g. ferrous implants, metallic clips, magnetically activated implanted devices such as cardiac pacemakers, etc).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08-04 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-12-19 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For all results participants=knees.
Groups:
- OtisMed® ShapeMatch® With Triathlon: Participants who underwent Total Knee Replacement (TKR) with the Stryker Triathlon® Total Knee System and OtisMed® ShapeMatch® Technology.
- Stryker Precision Knee Navigation: Participants who underwent Total Knee Replacement (TKR) with the Stryker Triathlon® Total Knee System guided by Stryker Precision Knee Navigation.
Period: Overall Study
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Started | 50 | 50
Completed | 49 | 50
Not Completed | 1 | 0
Not completed — Did not receive study intervention | 1 | 0

BASELINE CHARACTERISTICS:
Population: OtisMed Shapematch with Triathlon is the new intervention for component placement in total knee arthroplasty. This will be compared to the current standard (control) of Stryker Precision Knee Navigation.
Groups:
- Total: Total of all reporting groups
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (6.5) | 69.6 (7.5) | 70.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 24 | 24 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  New Zealand | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Oxford Knee Score
Description: To demonstrate, through calculation of Oxford Knee Score (OKS) post operatively, that total knee replacement (TKR) performed using the ShapeMatch® Cutting Guide provides improvement from preoperative levels of patient pain and function comparable to the improvement obtained with TKR performed using computer-assisted Navigation. Oxford Knee Scores will be calculated pre-operatively and at 6 weeks, 6 months, 12 months, 2 years and 5 years. The OKS is a participant completed 12 question form on activities of daily living that assess function and pain. Scores can range from 0 to 48 with lower scores indicating a poor outcome and higher scores indicating a more satisfactory joint outcome.
Time Frame: Preoperatively, 6-week, 6-months, 12 months, 2 years and 5 years postoperatively
Population: Shapematch: 49 had preoperative,48 had 6 week, 46 had 6 months, 48 had 12 month, 49 had 2 year and 47 had 5 year scores.
  Navigation: 50 had preoperative, 47 had 6 week, 46 had 6 months, 49 had 12 month, 50 had 2 years and 48 had 5 years scores.
  Participants=knees
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
units on a scale
  Oxford preoperative | 20.3 (5.7) | 21.1 (6.2)
  Oxford 6 weeks: number analyzed (Participants) | 48 | 47
  Oxford 6 weeks | 32.5 (6.8) | 32.8 (7.7)
  Oxford 6 months: number analyzed (Participants) | 46 | 46
  Oxford 6 months | 41.0 (4.8) | 38.2 (7.3)
  Oxford 12 months: number analyzed (Participants) | 48 | 49
  Oxford 12 months | 41.8 (6.1) | 43.0 (7.7)
  Oxford 2 years | 42.1 (6.1) | 41.1 (6.0)
  Oxford 5 years: number analyzed (Participants) | 47 | 48
  Oxford 5 years | 41.4 (7.2) | 41.7 (6.3)
Statistical Analysis 1: Comparison: Stryker Precision Knee Navigation; Improvement from preoperative to 6 weeks for the control cases; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: OtisMed® ShapeMatch® With Triathlon; Improvement from preoperative to 6 weeks for the Shapematch cases; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare improvement of OKS from preoperative to 6 weeks between both groups; Test type: Superiority; p = 0.0004, t-test, 2 sided
Statistical Analysis 4: Comparison: Stryker Precision Knee Navigation; Improvement from preoperative to 6 months for Control cases; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: OtisMed® ShapeMatch® With Triathlon; Improvement form preoperative to 6 months for Shapematch cases; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare improvement of OKS from preoperative to 6 months between both groups; Test type: Superiority; p = 0.3894, t-test, 2 sided
Statistical Analysis 7: Comparison: Stryker Precision Knee Navigation; Improvement from preoperative to 12 months for the Control cases; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: OtisMed® ShapeMatch® With Triathlon; Improvement from preoperative to 12 months for the Shapematch cases; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 9: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare improvement of OKS from preoperative to 12 months between both groups; Test type: Superiority; p = 0.4387, t-test, 2 sided; p-values from repeated ANOVA with change from preoperative variable/scores as dependent variable
Statistical Analysis 10: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare improvement of OKS from preoperative to 2 years between both groups; Test type: Superiority; p = 0.2610, t-test, 2 sided
Statistical Analysis 11: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare improvement of OKS from preoperative to 5 years between both groups; Test type: Superiority; p = 0.8458, t-test, 2 sided

2. Secondary Outcome: Cost Effectiveness: Total Duration of Operating Procedure (Anaesthetic Time and Skin-to-skin Incision Time)
Description: Skin to skin time is the time in minutes from initial skin incision to skin closure. Anaesthesia time is the time in minutes that anaesthesia administration is started to the time it is stopped. Data for anaesthesia time is not available due to an error on the original case report form that did not correctly capture anaesthesia time.
Time Frame: Intraoperative - participants were followed for the duration of the operation, an average of 1 hour and 50 minutes.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
minutes | 82.6 (26) | 92.2 (32)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare mean duration of surgery between both groups; Test type: Superiority; p = 0.10, t-test, 2 sided

3. Secondary Outcome: Cost Effectiveness: Wound Length
Description: To compare the cost-effectiveness and cost-utility of the procedure between the ShapeMatch® Cutting Guide group and the computer-assisted Navigation control group the surgical incision length is reported in mm.
Time Frame: Intraoperative - participants were followed for the duration of the operation, an average of 1 hour and 50 minutes.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
millimeters | 223 (29) | 233 (34)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare wound length between both groups; Test type: Superiority; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Cost Effectiveness: Cost of Consumable Items Used During Operating Procedure
Description: To compare the cost-effectiveness and cost-utility of the procedure between the ShapeMatch® Cutting Guide group and the computer-assisted Navigation control group. The data for the cost of consumable items used during the operating procedure is not available. Due to limited site resources, a decision was made not to collect this secondary outcome measure data.
Time Frame: Intraoperative - participants were followed for the duration of the operation, an average of 1 hour and 50 minutes.
Population: Cost effectiveness data is not available.
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cost Effectiveness: Length of Stay in Hospital
Description: To compare the cost-effectiveness and cost-utility of the procedure between the ShapeMatch® Cutting Guide group and the computer-assisted Navigation control group the length of stay in number of days spent in the hospital is reported..
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
days | 5.1 (3.0) | 4.2 (4.2)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare average length of hospital stay between both groups; Test type: Superiority; p = 0.07, t-test, 2 sided

6. Secondary Outcome: Cost Effectiveness: Quality-adjusted Life-years (QALYs) From EQ-5D-3L
Description: A quality-adjusted life-year (QALY) takes into account both the quantity and quality of life generated by healthcare interventions. It is the arithmetic product of life expectancy and a measure of the quality of the remaining life-years. A QALY places a weight on time in different health states. A year of perfect health is worth 1 and a year of less than perfect health is worth less than 1. Death is considered to be equivalent to 0; however,some health states may be considered worse than death and have negative scores.
Time Frame: 12 months
Population: Shapematch preoperative N=48, 12 month N=48.
  Navigation preoperative N=50, 12 month N-49.
Measure: Mean (Standard Deviation); unit: QALY life year
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 48 | 50
QALY life year
  Preoperative QALY | 0.507 (0.17) | 0.484 (0.21)
  12 Month QALY: number analyzed (Participants) | 48 | 49
  12 Month QALY | 0.895 (0.16) | 0.852 (0.19)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; Comparison of baseline differences; Test type: Superiority; p = 0.55, t-test, 2 sided; Mean Difference (Final Values) = -0.023
Statistical Analysis 2: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; Analysis of QALY between each instrument platform at 12-months; Test type: Superiority; p = 0.23, t-test, 2 sided; Mean Difference (Final Values) = -0.043

7. Secondary Outcome: Knee Pain
Description: Pain at rest and pain during mobilization was measured using a 10 centimeter Visual Analogue Scale (VAS). Participants are asked to indicate their level of pain with 0 being no pain and 10 being the worst pain.
Time Frame: Preoperatively, 6-week, 6-months,12 months, 2 years and 5 years postoperatively
Population: Patients did not complete CRF to protocol in some instances, resulting in exclusion/missing data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OtisMed® ShapeMatch® With Triathlon: Participants randomised to the Intervention Group will undergo Total Knee Replacement (TKR) with the Stryker Triathlon® Total Knee System and OtisMed® ShapeMatch® Technology with the goal of kinematic alignment (re-aligning the limb to its pre-disease kinematic alignment).
  OtisMed® ShapeMatch® Technology: The appropriate Stryker ShapeMatch® Cutting Guides will be used to guide the surgeons bone resections. The surgeon will implant the knee prostheses following the surgical protocol for Triathlon® Knee System with OtisMed® ShapeMatch® Technology
  Total Knee Replacement
  Stryker Triathlon® Total Knee System: Prosthetic components to be implanted including
  * Triathlon® Cruciate Retaining (CR) Total Knee System (cemented), including Femoral Component and Primary Tibial Baseplate;
  * Triathlon® Cruciate Substituting (CS) X3® polyethylene insert;
  * Triathlon® X3 Patella (asymmetric) - treated selectively by surgeon.
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
score on a scale
  Pre-op Pain at Rest | 4.36 (2.03) | 4.20 (2.48)
  Pre-op Pain at Mobilisation | 5.78 (2.32) | 6.01 (2.49)
  6-week Pain at Rest: number analyzed (Participants) | 48 | 47
  6-week Pain at Rest | 1.95 (1.93) | 1.79 (2.01)
  6-week Pain at Mobilisation: number analyzed (Participants) | 48 | 47
  6-week Pain at Mobilisation | 2.51 (2.11) | 2.49 (2.00)
  6-month Pain at Rest: number analyzed (Participants) | 46 | 45
  6-month Pain at Rest | 0.97 (1.78) | 1.20 (2.04)
  6-month Pain at Mobilisation: number analyzed (Participants) | 46 | 45
  6-month Pain at Mobilisation | 1.15 (1.97) | 1.50 (2.38)
  1-year Pain at Rest: number analyzed (Participants) | 46 | 49
  1-year Pain at Rest | 0.53 (1.35) | 0.84 (1.63)
  1-year Pain at Mobilisation: number analyzed (Participants) | 46 | 48
  1-year Pain at Mobilisation | 0.79 (1.83) | 1.35 (2.3)
  2-year Pain at Rest: number analyzed (Participants) | 48 | 50
  2-year Pain at Rest | 0.67 (0.94) | 1.00 (1.72)
  2-year Pain at Mobilisation: number analyzed (Participants) | 48 | 50
  2-year Pain at Mobilisation | 1.14 (1.35) | 1.31 (1.84)
  5-year Pain at Rest: number analyzed (Participants) | 47 | 48
  5-year Pain at Rest | 0.84 (1.56) | 0.63 (1.07)
  5-year Pain at Mobilisation: number analyzed (Participants) | 47 | 48
  5-year Pain at Mobilisation | 1.21 (1.64) | 1.17 (2.06)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS rest preoperatively between both groups; Test type: Equivalence — To determine equivalence in baseline characteristics between the control and intervention group; p = 0.7240, t-test, 2 sided
Statistical Analysis 2: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS mobilisation preoperatively between both groups; Test type: Equivalence — To determine equivalence in baseline characteristics between the control and intervention group; p = 0.7545, t-test, 2 sided
Statistical Analysis 3: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS rest at 6 weeks between both groups; Test type: Non-Inferiority — Precision Knee Navigation is the current standard of care and is the control against the newer intervention of OtisMed® ShapeMatch® with Triathlon; p = 0.6921, t-test, 2 sided
Statistical Analysis 4: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS mobilisation at 6 weeks between both groups; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 3]; p = 0.9601, t-test, 2 sided
Statistical Analysis 5: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS rest at 6 months between both groups; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 3]; p = 0.0697, t-test, 2 sided
Statistical Analysis 6: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS mobilisation at 6 months between both groups; Test type: Equivalence — [test comment as in outcome 7, analysis 3]; p = 0.0342, t-test, 2 sided
Statistical Analysis 7: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS rest at 12 months between both groups; Test type: Equivalence — [test comment as in outcome 7, analysis 3]; p = 0.3487, t-test, 2 sided
Statistical Analysis 8: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS mobilisation at 1 year between both groups; Test type: Equivalence — [test comment as in outcome 7, analysis 3]; p = 0.2201, t-test, 2 sided
Statistical Analysis 9: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS rest at 2 years between both groups; Test type: Equivalence — [test comment as in outcome 7, analysis 3]; p = 0.2291, t-test, 2 sided
Statistical Analysis 10: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS mobilisation at 2 years between both groups; Test type: Equivalence — [test comment as in outcome 7, analysis 3]; p = 0.6436, t-test, 2 sided
Statistical Analysis 11: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS rest at 5 years between both groups; Test type: Equivalence — [test comment as in outcome 7, analysis 3]; p = 0.4344, t-test, 2 sided
Statistical Analysis 12: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare VAS mobilisation at 5 years between both groups; Test type: Equivalence — [test comment as in outcome 7, analysis 3]; p = 0.8732, t-test, 2 sided

8. Secondary Outcome: The Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: The WOMAC is completed by the participant and measures five items for pain (score range 0-100), two for stiffness (score range 0-100), and 17 for functional limitation (score range 0-100). The total score is the sum of these three categories.
Time Frame: Preoperatively, 6-week, 6-months,12 months, 2 years and 5 years postoperatively
Population: Patients did not complete CRF to protocol in some instances, resulting in exclusion/missing data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
score on a scale
  Pre-op | 50.05 (13.07) | 50.36 (14.91)
  6-week: number analyzed (Participants) | 48 | 47
  6-week | 74.74 (11.75) | 73.06 (17.61)
  6-month: number analyzed (Participants) | 46 | 46
  6-month | 87.89 (9.73) | 81.79 (15.94)
  1-year: number analyzed (Participants) | 48 | 49
  1-year | 90.86 (11.14) | 86.79 (14.93)
  2-year | 88.36 (13.60) | 85.46 (16.79)
  5-year: number analyzed (Participants) | 47 | 48
  5-year | 86.13 (15.49) | 89.14 (15.11)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare WOMAC preoperatively between both groups; Test type: Superiority; p = 0.911, t-test, 2 sided
Statistical Analysis 2: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare WOMAC at 6-weeks between both groups; Test type: Superiority; p = 0.588, t-test, 2 sided
Statistical Analysis 3: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare WOMAC at 6-months between both groups; Test type: Superiority; p = 0.030, t-test, 2 sided
Statistical Analysis 4: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare WOMAC at 1-year between both groups; Test type: Superiority; p = 0.131, t-test, 2 sided
Statistical Analysis 5: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare WOMAC at 2-years between both groups; Test type: Superiority; p = 0.347, t-test, 2 sided
Statistical Analysis 6: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare WOMAC at 5-years between both groups; Test type: Superiority; p = 0.341, t-test, 2 sided

9. Secondary Outcome: Health-related Quality of Life (EQ-5D-3L)
Description: The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The participant is asked to indicate his/her health state by indicating the most appropriate level for each of the 5 dimensions. Responses may be converted into a single summary index by applying a formula that essentially attaches values (also called weights) to each of the levels in each dimension. The index can be calculated by deducting the appropriate weights from 1= the value for full health.
  The EQ VAS records the participant's self-rated health on a vertical, visual analogue scale where the endpoints are labelled from 100 ='Best imaginable health state' to 0= 'Worst imaginable health state'.
Time Frame: Preoperatively, 6-week, 6-month and 12 month visits, 2 years and 5 years
Population: Patients did not complete CRF to protocol in some instances, resulting in exclusion/missing data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
score on a scale
  Pre-op EQ-5D Index: number analyzed (Participants) | 48 | 50
  Pre-op EQ-5D Index | 0.51 (0.17) | 0.48 (0.21)
  Pre-op EQ-5D VAS | 71.43 (18.11) | 75.66 (14.28)
  6-week EQ-5D Index: number analyzed (Participants) | 48 | 46
  6-week EQ-5D Index | 0.67 (0.14) | 0.68 (0.18)
  6-week EQ-5D VAS: number analyzed (Participants) | 48 | 47
  6-week EQ-5D VAS | 79.38 (13.58) | 80.28 (19.41)
  6-month EQ-5D Index: number analyzed (Participants) | 46 | 45
  6-month EQ-5D Index | 0.82 (0.18) | 0.78 (0.2)
  6-month EQ-5D VAS: number analyzed (Participants) | 45 | 45
  6-month EQ-5D VAS | 86.00 (13.86) | 84.04 (14.52)
  1-year EQ-5D Index: number analyzed (Participants) | 48 | 49
  1-year EQ-5D Index | 0.89 (0.16) | 0.84 (0.20)
  1-year EQ-5D VAS: number analyzed (Participants) | 48 | 47
  1-year EQ-5D VAS | 85.48 (12.46) | 85.91 (12.22)
  2-year EQ-5D Index | 0.77 (0.30) | 0.70 (0.30)
  2-year EQ-5D VAS | 81.80 (18.57) | 84.70 (11.63)
  5-year EQ-5D Index: number analyzed (Participants) | 47 | 47
  5-year EQ-5D Index | 0.82 (0.20) | 0.86 (0.18)
  5-year EQ-5D VAS: number analyzed (Participants) | 47 | 48
  5-year EQ-5D VAS | 78.21 (16.51) | 78.58 (17.02)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D index preoperatively between both groups; Test type: Superiority; p = 0.452, t-test, 2 sided
Statistical Analysis 2: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D VAS preoperatively between both groups; Test type: Superiority; p = 0.201, t-test, 2 sided
Statistical Analysis 3: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D index at 6-weeks between both groups; Test type: Superiority; p = 0.741, t-test, 2 sided
Statistical Analysis 4: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D VAS at 6-weeks between both groups; Test type: Superiority; p = 0.794, t-test, 2 sided
Statistical Analysis 5: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D index at 6-months between both groups; Test type: Superiority; p = 0.232, t-test, 2 sided
Statistical Analysis 6: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D VAS at 6-months between both groups; Test type: Superiority; p = 0.513, t-test, 2 sided
Statistical Analysis 7: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D index at 1-year between both groups; Test type: Superiority; p = 0.180, t-test, 2 sided
Statistical Analysis 8: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D VAS at 1-year between both groups; Test type: Superiority; p = 0.864, t-test, 2 sided
Statistical Analysis 9: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D index at 2-year between both groups; Test type: Superiority; p = 0.223, t-test, 2 sided
Statistical Analysis 10: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D VAS at 2-year between both groups; Test type: Superiority; p = 0.355, t-test, 2 sided
Statistical Analysis 11: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D index at 5-year between both groups; Test type: Superiority; p = 0.314, t-test, 2 sided
Statistical Analysis 12: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare EQ-5D VAS at 5-year between both groups; Test type: Superiority; p = 0.914, t-test, 2 sided

10. Secondary Outcome: The Forgotten Joint Score (FJS-12)
Description: The Forgotten Joint Score (FJS) is a 12 question form that asks the patient their level of awareness of their artificial joint in 12 scenarios commonly encountered in daily life. Scores can range from 0 to 100 with a higher score indicating a better outcome (high degree of forgetting the joint in everyday life).
Time Frame: 6 week, 6 month, 12 month , 2 years and 5 years visits
Population: Patients did not complete CRF to protocol in some instances, resulting in exclusion/missing data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
score on a scale
  6 week: number analyzed (Participants) | 46 | 46
  6 week | 58.12 (25.53) | 57.21 (29.32)
  6 month: number analyzed (Participants) | 48 | 46
  6 month | 60.47 (29.57) | 59.96 (28.27)
  12 month: number analyzed (Participants) | 47 | 49
  12 month | 62.47 (28.99) | 62.01 (24.84)
  2 year | 69.21 (25.93) | 66.22 (25.54)
  5 year: number analyzed (Participants) | 47 | 48
  5 year | 68.04 (28.824) | 74.12 (23.38)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare FJS at 6-weeks between both groups; Test type: Superiority; p = 0.523, t-test, 2 sided
Statistical Analysis 2: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare FJS at 6-months between both groups; Test type: Superiority; p = 0.932, t-test, 2 sided
Statistical Analysis 3: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare FJS at 1-year between both groups; Test type: Superiority; p = 0.934, t-test, 2 sided
Statistical Analysis 4: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare FJS at 2-year between both groups; Test type: Superiority; p = 0.566, t-test, 2 sided
Statistical Analysis 5: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare FJS at 5-year between both groups; Test type: Superiority; p = 0.263, t-test, 2 sided

11. Secondary Outcome: The International Knee Society Score (IKSS)
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a minimum score of 0 to a maximum of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: Preoperatively, 6-week, 6-months,12 months, 2 years and 5 years postoperatively
Population: Patients did not complete CRF to protocol in some instances, resulting in exclusion/missing data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
score on a scale
  Pre-op IKSS Pain: number analyzed (Participants) | 44 | 46
  Pre-op IKSS Pain | 40.20 (15.87) | 37.33 (14.82)
  Pre-op IKSS Function: number analyzed (Participants) | 48 | 50
  Pre-op IKSS Function | 54.06 (15.70) | 55.50 (14.82)
  Pre-op Range of Motion: number analyzed (Participants) | 44 | 47
  Pre-op Range of Motion | 118.07 (11.27) | 116.17 (15.51)
  6 week IKSS Pain: number analyzed (Participants) | 41 | 37
  6 week IKSS Pain | 63.02 (15.37) | 58.30 (18.28)
  6 week IKSS Function: number analyzed (Participants) | 48 | 47
  6 week IKSS Function | 63.33 (16.90) | 64.26 (22.26)
  6 week Range of Motion: number analyzed (Participants) | 44 | 46
  6 week Range of Motion | 108.64 (17.58) | 107.28 (14.99)
  6 month IKSS Pain: number analyzed (Participants) | 34 | 35
  6 month IKSS Pain | 76.32 (12.72) | 68.77 (18.81)
  6 month IKSS Function: number analyzed (Participants) | 46 | 46
  6 month IKSS Function | 82.17 (17.72) | 76.85 (21.30)
  6 month Range of Motion: number analyzed (Participants) | 46 | 43
  6 month Range of Motion | 117.24 (13.31) | 113.09 (21.31)
  12 month IKSS Pain: number analyzed (Participants) | 47 | 45
  12 month IKSS Pain | 76.96 (14.65) | 73.29 (15.08)
  12 month IKSS Function: number analyzed (Participants) | 48 | 49
  12 month IKSS Function | 83.96 (17.38) | 80.82 (20.22)
  12 month Range of Motion: number analyzed (Participants) | 48 | 47
  12 month Range of Motion | 118.19 (12.69) | 116.57 (12.11)
  2 year IKSS Pain: number analyzed (Participants) | 33 | 31
  2 year IKSS Pain | 73.67 (9.92) | 70.10 (16.32)
  2 year IKSS Function: number analyzed (Participants) | 49 | 48
  2 year IKSS Function | 83.06 (17.94) | 80.52 (23.00)
  2 year Range of Motion: number analyzed (Participants) | 48 | 48
  2 year Range of Motion | 119.19 (11.91) | 117.63 (15.20)
  5 year IKSS Pain: number analyzed (Participants) | 38 | 42
  5 year IKSS Pain | 73.26 (12.19) | 74.71 (8.95)
  5 year IKSS Function: number analyzed (Participants) | 47 | 47
  5 year IKSS Function | 80.96 (18.41) | 85.96 (16.64)
  5 year Range of Motion: number analyzed (Participants) | 42 | 46
  5 year Range of Motion | 122.24 (6.69) | 120.43 (9.16)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Pain preoperatively between both groups; Test type: Superiority; p = 0.3768, t-test, 2 sided
Statistical Analysis 2: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Function preoperatively between both groups; Test type: Superiority; p = 0.6425, t-test, 2 sided
Statistical Analysis 3: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS ROM preoperatively between both groups; Test type: Superiority; p = 0.5041, t-test, 2 sided
Statistical Analysis 4: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Pain at 6-weeks between both groups; Test type: Superiority; p = 0.2230, t-test, 2 sided
Statistical Analysis 5: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Function at 6-weeks between both groups; Test type: Superiority; p = 0.8209, t-test, 2 sided
Statistical Analysis 6: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS ROM at 6-weeks between both groups; Test type: Superiority; p = 0.6958, t-test, 2 sided
Statistical Analysis 7: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Pain at 6-months between both groups; Test type: Superiority; p = 0.0548, t-test, 2 sided
Statistical Analysis 8: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Function at 6-months between both groups; Test type: Superiority; p = 0.1958, t-test, 2 sided
Statistical Analysis 9: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS ROM at 6-months between both groups; Test type: Superiority; p = 0.2786, t-test, 2 sided
Statistical Analysis 10: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Pain at 1-year between both groups; Test type: Superiority; p = 0.2399, t-test, 2 sided
Statistical Analysis 11: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Function at 1-year between both groups; Test type: Superiority; p = 0.4135, t-test, 2 sided
Statistical Analysis 12: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS ROM at 1-year between both groups; Test type: Superiority; p = 0.5278, t-test, 2 sided
Statistical Analysis 13: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Pain at 2-year between both groups; Test type: Superiority; p = 0.2992, t-test, 2 sided
Statistical Analysis 14: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Function at 2-year between both groups; Test type: Superiority; p = 0.5462, t-test, 2 sided
Statistical Analysis 15: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS ROM at 2-year between both groups; Test type: Superiority; p = 0.5765, t-test, 2 sided
Statistical Analysis 16: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Pain at 5-year between both groups; Test type: Superiority; p = 0.5493, t-test, 2 sided
Statistical Analysis 17: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS Function at 5-year between both groups; Test type: Superiority; p = 0.1705, t-test, 2 sided
Statistical Analysis 18: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; To compare IKSS ROM at 5-year between both groups; Test type: Superiority; p = 0.2918, t-test, 2 sided

12. Secondary Outcome: Perth CT Protocol
Description: The Perth CT protocol is a comprehensive assessment of total knee replacement (TKR) component position and orientation. The alignment of the TKR components is measured against the mechanical axis and the transepicondylar axis of the lower extremity. The posted data represents the mean angle between the femoral component and mechanical axis of the femur, the angle between tibial component and mechanical axis of the tibia, the tibial component slope relative to the sagittal mechanical axis, and the femoral component rotation relative to surgical epicondylar axis (positive value=external rotation). For all degree values posted a positive (+) value= valgus and a negative (-) value = varus.
Time Frame: 3 months
Population: Participants=knees
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
Number analyzed (Participants) | 49 | 50
degrees
  Coronal mechanical axis:hip knee ankle angle | -0.4 (3.5) | -0.7 (2.0)
  Coronal angle fem comp and mech axis femur | 2.0 (2.6) | 0.6 (1.6)
  Coronal angle tibial comp and mech axis tibia | -2.8 (3.1) | -0.7 (1.9)
  Sagital tibial component slope | 3.6 (2.5) | 1.3 (2.4)
  Femcomp rotationrelative to surg epicond axis+=ER | -0.5 (2.5) | 1.5 (2.5)
Statistical Analysis 1: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; Comparison of coronal mechanical axis:hip knee ankle angle between both groups; Test type: Other; p = 0.6, t-test, 2 sided
Statistical Analysis 2: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; Comparison of coronal angle fem comp and mech axis femur between both groups; Test type: Other; p = 0.002, t-test, 2 sided
Statistical Analysis 3: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; Comparison of coronal angle tibial comp and mech axis tibia between both groups; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; Comparison of sagital tibial component slope between both groups; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: OtisMed® ShapeMatch® With Triathlon vs Stryker Precision Knee Navigation; Comparison of Fem comp rotation relative to surg epicond axis+=ER between both groups; Test type: Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 5-years
Description: Elective procedures not included.e.g.non-study joint replacement/revision, rotator cuff repair,carpal tunnel release,cataract,intra-ocular & bunion procedures,total shoulder repair,laminectomy,microdiscectomy,breast reduction,cervical spine fusion,& mid/flat-foot surgery.Industry standard AE terms not used;specific AE terms not used for all AEs.
Arm/Group | OtisMed® ShapeMatch® With Triathlon | Stryker Precision Knee Navigation
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 39/49 | 38/50
Other Adverse Events (participants affected / at risk) | 24/49 | 25/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OtisMed® ShapeMatch® With Triathlon (N=49) | Stryker Precision Knee Navigation (N=50)
Non-operative site (Cardiac disorders) | 5 (6) | 4 (5)
Non-operative site (Gastrointestinal disorders) | 4 (5) | 10 (11)
Non-operative site (General disorders) | 3 (3) | 3 (6)
Non-operative site (Hepatobiliary disorders) | 3 (3) | 2 (2)
Operative site (Infections and infestations) | 1 (1) | 3 (3)
Non-operative site (Musculoskeletal and connective tissue disorders) | 21 (26) | 21 (33)
Operative site (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Non-operative site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Non-operative site (Psychiatric disorders) | 2 (2) | 0 (0)
Non-operative site (Renal and urinary disorders) | 2 (2) | 3 (4)
Non-operative site (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 8 (8)
Non-operative site (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Non-operative site (Vascular disorders) | 4 (5) | 3 (4)
Non-operative site (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Non-operative site (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Non-operative site (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Non-operative site (Congenital, familial and genetic disorders) | 0 (0) | 0 (0)
Non-operative site (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Non-operative site (Endocrine disorders) | 0 (0) | 0 (0)
Non-operative site (Eye disorders) | 4 (5) | 4 (4)
Non-operative site (Immune system disorders) | 0 (0) | 0 (0)
Non-operative site (Infections and infestations) | 5 (5) | 9 (13)
Operative site (Investigations) | 1 (1) | 1 (1)
Non-operative site (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Non-operative side (Nervous system disorders) | 0 (0) | 2 (3)
Non-operative side (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Non-operative side (Product Issues) | 0 (0) | 0 (0)
Non-operative site (Social circumstances) | 0 (0) | 0 (0)
Operative site (Surgical and medical procedures) | 3 (3) | 4 (7)
Non-operative site (Surgical and medical procedures) | 25 (35) | 28 (42)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OtisMed® ShapeMatch® With Triathlon (N=49) | Stryker Precision Knee Navigation (N=50)
Operative site (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
Non-operative site (Eye disorders) | 3 (3) | 2 (2)
Non-operative site (Gastrointestinal disorders) | 6 (7) | 2 (3)
Non-operative site (General disorders) | 0 (0) | 3 (3)
Non-operative site (Infections and infestations) | 2 (3) | 5 (6)
Non-operative site (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Operative site (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Non-operative site (Musculoskeletal and connective tissue disorders) | 8 (12) | 10 (14)
Operative site (Product Issues) | 6 (6) | 0 (0)
Non-operative site (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Non-operative site (Surgical and medical procedures) | 7 (9) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discloser must give at least 40 days notice to Sponsor including a copy of the proposed publication. The Sponsor can then provide comments (which Discloser is not bound to follow), request delay of publication by no more than 120 days to allow for Sponsor to protect its intellectual property, or request that the Discloser remove certain proprietary or confidential information from the study (other than the results of the study).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT02527148/Prot_SAP_000.pdf